CLINICAL TRIAL: NCT03386526
Title: A Phase I Study of the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of APG-1387 as a Single Agent or in Combination With Systemic Anti-Cancer Agents in Patients With Advanced Solid Tumors or Hematologic Malignancies
Brief Title: APG-1387 in Patients With Advanced Solid Tumors or Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG-1387-US-001
Record Dates: First submitted 2017-12-13; First posted 2017-12-29 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumors or Hematologic Malignancies
Keywords: IAP inhibitor
MeSH Terms: conditions — Hematologic Neoplasms | interventions — APG-1387; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APG-1387 for Injection (Experimental): APG-1387 will be explored sequentially using a standard 3+3 escalation scheme at the dose escalation phase and up to 20 patient per group at the dose expansion phase.
  Interventions: Drug: APG-1387 for Injection

INTERVENTIONS:
Drug: APG-1387 for Injection — Multiple dose cohorts, 30 minute IV infusion, once weekly for 3 weeks of a 21-day cycle

SUMMARY:
APG-1387 is a potent, bivalent small-molecule Inhibitor of Apoptosis Protein (IAP) antagonist. APG-1387 has shown strong dose- and schedule-dependent antitumor activities in multiple human cancer xenograft models, APG-1387 also demonstrates its synergistic effect in combination with immune checkpoint inhibitor anti-PD-1 antibody, and such a combinatory effect was further enhanced by chemotherapeutic agent. A total of 35 patients with advanced solid tumors or lymphomas have been treated with APG-1387 in two Phase I dose-escalation studies in Australia and in China. Ten dose levels have been tested ranging from 0.3 mg to 45 mg in these two studies. Based on the preliminary results, APG-1387 is well-tolerated at the dose levels evaluated to date. APG-1387 is intended for the treatment of patients with advanced solid tumors and hematologic malignancies. After establishing the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and/or recommended phase 2 dose (RP2D), several Ib /II studies will be implemented accordingly to further access the antitumor effects of APG-1387 in combination with either pembrolizumab or the chemotherapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid tumor or hematological malignancies
2. Life expectancy ≥ 3 months
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
4. Corrected QT interval (QTc) ≤ 450 ms in males, and ≤ 470 ms in females
5. Adequate hematologic function
6. International normalized ratio (INR), prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5 x upper limit of normal (ULN)
7. Adequate renal and liver function
8. Willingness to use contraception
9. Ability to understand and willingness to sign a written informed consent form
10. Willingness and ability to comply with study procedures and follow-up examination
11. Have provided tissue for biomarker analysis from a newly or recently-obtained biopsy of a tumor lesion not previously irradiated

Exclusion Criteria:

1. Received chemotherapy within 21 days (42 days for nitrosoureas or mitomycin C) prior to entering the study
2. Received hormonal, biologic (< 2 half-lives), small molecule targeted therapies or other anti-cancer therapy within 21 days of study entry
3. Radiation or surgery within 14 days of study entry, thoracic radiation within 28 days of study entry
4. Has known active central nervous (CNS) metastases and/or carcinomatous meningitis. Patients who have received prior radiotherapy for previous brain metastasis must have discontinued steroids for 14 days prior to study entry and be clinically stable
5. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to ≤ Grade 1 except alopecia
6. Requirement for corticosteroid treatment, with the exception of megestrol, local use of steroid
7. Use of therapeutic anticoagulants
8. International normalized ratio (INR) or activated partial thromboplastin time (APTT) ≥ 1.5 x ULN
9. Concurrent treatment with an investigational agent or device within 28 days prior to the first dose of therapy
10. Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry
11. Neurologic instability per clinical evaluation due to tumor involvement of the central nervous system (CNS)
12. History of Bell's palsy
13. Active rheumatoid arthritis (RA), active inflammatory bowel disease, chronic infections, or any other disease or condition associated with chronic inflammation
14. Active infection requiring systemic antibiotic/ antifungal medication
15. Known or suspected Wilson's Disease
16. Prior treatment with IAP inhibitors
17. History of hypersensitivity to paclitaxel, or any therapeutic antibody
18. Has an active autoimmune disease, or a documented history of autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents
19. Is on chronic systemic steroid therapy
20. Has received a live vaccine within 30 days prior to first dose
21. Has had an allogeneic tissue/solid organ transplant, prior stem cell or bone marrow transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 18-24 months
  Patients with APG-1387 treatment related adverse events (AE), serious adverse events (SAE) will be assessed according NCI CTCAE Version 4.03

SECONDARY OUTCOMES:
Anti-tumor effects of APG-1387 as a single agent | 18-24 months
  Response will be evaluated every 2 cycles (8 weeks), according to the revised RECIST Guideline, Version 1.1 or the Revised Response Criteria for Malignant Lymphoma
Pharmacokinetic evaluation | 18-24 months
  Maximum plasma concentration (Cmax) will be assessed in the patients treated with APG-1387
Anti-tumor effects of APG-1387 in combination with pembrolizumab or combination with paclitaxel and carboplatin in patients with advanced solid tumors | 18-24 months
  Response will be evaluated every 2 cycles (8 weeks), according to the revised RECIST Guideline, Version 1.1 or the Revised Response Criteria for Malignant Lymphoma
Preliminary biomarker assessment | 18-24 months
  Tumor biopsy and peripheral blood sample at baseline and 15-21 days after administration of APG-1387 alone or in combination with systemic anti-cancer therapy
Pharmacokinetic evaluation | 18-24 months
  Area under the plasma concentration versus time curve (AUC) of APG-1387 will be assessed on patients treated with APG-1387

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - START Midwest, Grand Rapids, Michigan
  - The START Center for Cancer Care, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan W, Luo Q, Liang E, Shi M, Sun J, Shen H, Lu Z, Zhang L, Yan X, Yuan L, Zhou S, Yi H, Zhai Y, Qiu MZ, Yang D. Synergistic effects of Smac mimetic APG-1387 with anti-PD-1 antibody are attributed to increased CD3 + NK1.1 + cell recruitment secondary to induction of cytokines from tumor cells. Cancer Cell Int. 2024 May 24;24(1):181. doi: 10.1186/s12935-024-03373-7. PMID 38790057